CLINICAL TRIAL: NCT04481971
Title: Comparative Evaluation of the Effectiveness of Premedication With Two Different Single Doses of Prednisolone on Inter-appointment Pain in Symptomatic Patients With Irreversible Pulpitis: a Double-blind Randomized Controlled Clinical Trial
Brief Title: A Comparison of Two Different Single Doses of Prednisolone on Endodontic Inter-appointment Pain
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Sara Alsubait, Associate Professor, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-20-4818
Record Dates: First submitted 2020-07-12; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Endodontics; Pain
MeSH Terms: conditions — Pain | interventions — Prednisolone; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 40 mg (Experimental)
  Interventions: Drug: Prednisolone
- 20 mg (Experimental)
  Interventions: Drug: Prednisolone
- Placebo (Placebo Comparator)
  Interventions: Drug: lactose in capsules gelatin

INTERVENTIONS:
Drug: Prednisolone — Tablets
  Arms: 20 mg; 40 mg
Drug: lactose in capsules gelatin — Tablets
  Arms: Placebo

SUMMARY:
The purpose of this prospective randomized, double-blind, placebo-controlled study is to compare the efficiency of 2 different single doses of pre-operative oral prednisolone (20 & 40 mg) for the control of inter-appointment endodontic pain in patients diagnosed with symptomatic irreversible pulpitis. The tested null hypothesis is that there is no difference in pain relief between the two doses.

Seventy-two patients presented for treatment at Dental University Hospital will be selected. The inclusion criteria are systemically healthy patients (ASA classification I or II), with no contraindications to corticosteroids (osteoporosis, systemic fungal infections, poorly controlled insulin-dependent diabetes mellitus, ocular herpes simplex, primary glaucoma, allergy to corticosteroids, ulcerative colitis, a compromised immune status, and major psychosis). Patients under 18 years, pregnant or breast-feeding, took an analgesic agent within the last 6 hours, those with un-restorable teeth, teeth with periodontal disease will be excluded. Patients having mandibular molars with symptomatic irreversible pulpitis with normal periapical area and moderate-severe preoperative pain (i.e. ≥ 34 mm on a visual analog scale (VAS)) will be included.

Subjects will be randomly divided into 3 groups, namely placebo (control), 20 mg prednisolone and 40 mg prednisolone according to a computerized random numbers. Each participant will receive a single oral dose of either formulation (drug or placebo) 30 minutes before starting endodontic treatment. All medications will be placed in identical containers and will be coded; thus, both the operator and the patients will be blinded to the type of medication. Endodontic treatment will be performed and canals will be instrumented to a minimum of size 30, .04 taper following the standardized protocol. Postoperative pain will be assessed by using a visual analogue scale at 4, 12, 24 and 48 hours after initiation of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients (ASA classification I or II), with no contraindications to corticosteroids (osteoporosis, systemic fungal infections, poorly controlled insulin- dependent diabetes mellitus, ocular herpes simplex, primary glaucoma, allergy to corticosteroids, ulcerative colitis, a compromised immune status, and major psychosis).

Exclusion Criteria:

* Patients under 18 years, pregnant or breast-feeding, took an analgesic agent within the last 6 hours, those with un-restorable teeth, teeth with periodontal disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-08-09 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in post-operative pain | Change from baseline pain and pain at 4, 12, 24, and 48 hours after initiation of therapy
  Questionnaire (visual analogue scale)